CLINICAL TRIAL: NCT03579394
Title: CHRONO - Retarded Surgery Following Neoadjuvant Chemotherapy in Advanced Ovarian Cancer
Brief Title: Retarded Surgery Following Neoadjuvant Chemotherapy in Advanced Ovarian Cancer
Acronym: CHRONO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: ARCAGY/ GINECO GROUP (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GINECO-CHIR101
Record Dates: First submitted 2018-05-31; First posted 2018-07-06 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Ovarian Cancer Stage IV; Ovarian Cancer Stage IIIC; Ovarian Cancer Stage IIIb
Keywords: ovarian cancer; retarded surgery; neoadjuvant chemotherapy
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Interval Debulking Surgery (IDS) (Active Comparator): Complete surgery after 3 courses of neoadjuvant chemotherapy (NACT)
  Interventions: Procedure: Standard IDS (Interval Debulking Surgery)
- Retarded Interval Debulking Surgery (IDS) (Experimental): Complete surgery after 6 courses of neoadjuvant chemotherapy (NACT)
  Interventions: Procedure: Retarded IDS (Interval Debulking Surgery)

INTERVENTIONS:
Procedure: Retarded IDS (Interval Debulking Surgery) — Patient will receive 6 courses of i.v carboplatine and paclitaxel every 3 weeks followed by IDS (Interval Debulking Surgery) within 6 weeks from C6D1. After surgery patient will undergo 2 more courses of carboplatine and paclitaxel chemotherapy
  Treatment accepted :
  Paclitaxel and carboplatin could will be administred according to the site practice and Saint-Paul-de-Vence recommendation (Joly et al, 2017):
  * paclitaxel 175 mg/m² + carboplatin AUC 5-6, D1=D21 or
  * paclitaxel 80 mg/m² at J1-J8-J15 + carboplatin AUC 5-6, D1=D21 or
  * paclitaxel 60 mg/m² D1-D8-D15 + carboplatin AUC2 D1-D8-D15, D1= D21
  * Adjuvant therapy and maintenance (optional)according to national recommendations (Saint Paul de Vence)
  Arms: Retarded Interval Debulking Surgery (IDS)
Procedure: Standard IDS (Interval Debulking Surgery) — Patient will receive 3 courses of i.v carboplatine and paclitaxel every 3 weeks followed by IDS (Interval Debulking Surgery) within 6 weeks from C3D1. After surgery patient will undergo 5 more courses of carboplatine and paclitaxel chemotherapy.
  Treatment accepted :
  Paclitaxel and carboplatin could will be administred according to the site practice and Saint-Paul-de-Vence recommendation (Joly et al, 2017):
  * paclitaxel 175 mg/m² + carboplatin AUC 5-6, D1=D21 or
  * paclitaxel 80 mg/m² at J1-J8-J15 + carboplatin AUC 5-6, D1=D21 or
  * paclitaxel 60 mg/m² D1-D8-D15 + carboplatin AUC2 D1-D8-D15, D1= D21
  * Adjuvant therapy and maintenance (optional)according to national recommendations (Saint Paul de Vence)
  Arms: Interval Debulking Surgery (IDS)

SUMMARY:
The aim of CHRONO trial is to compare the DFS when surgery is performed after 3 courses of NACT, or after 6 courses of NACT, in a prospective multi institutional randomized setting,considering only patients initially unsuitable for primary surgery.

ELIGIBILITY:
Inclusion Criteria:

1. Female patients ≥18 years.
2. Histologically confirmed epithelial ovarian cancer, fallopian tube carcinoma or primary peritoneal carcinoma, high grade serous or endometrioïd, with the exception of mucinous, clear cell and carcinosarcoma histologies.
3. Performance status < 2 (see Appendix 2).
4. Documented International Federation of Gynecologic Oncology (FIGO 2014, Appendix 1) stage IIIB-IIIC-IVa unsuitable for complete primary cytoreductive surgery (confirmed by open laparoscopy or by laparotomy [not mandatory for stage IVA]).
5. Patient must be judged resectable after 3 courses of Neoadjuvant chemotherapy
6. Adequate bone marrow, liver and renal function to receive chemotherapy and subsequently to undergo surgery:

   * White blood cells (WBC) >3x109/L, absolute neutrophil count (ANC) ≥1,5x109/L, platelets (PLT)

     ≥100x109/L, hemoglobin (Hb) ≥9 g/dL,
   * Serum creatinine <1.25 x upper normal limit (UNL) or creatinine clearance ≥ 30 mL/min according to Cockroft-Gault formula or to local lab measurement, serum bilirubin <1.25 x UNL, AST(SGOT) and ALT(SGPT) <2.5 x UNL.
7. Signed informed consent obtained prior to any study-specific procedures.
8. Patient affiliated to, or a beneficiary of, a social security category

Exclusion Criteria:

1. Mucinous, clear cell , carcinosarcoma and low grade serous carcinomahistologies.
2. Synchronous or previous other malignancies within 3 years prior to starting study treatment, with the exception of adequately treated non-melanomatous skin cancer or carcinoma in situ (of the cervix or breast or other sites).
3. Patients with brain metastases, seizure not controlled with standard medical therapy, or history of cerebrovascular accident (CVA, stroke) or transient ischemic attack (TIA) or subarachnoid hemorrhage before 6 months from the enrollment on this study.
4. Any other concurrent medical conditions contraindicating surgery or chemotherapy that could compromise the adherence to the protocol (including but not limited to impaired cardiac function or clinically significant cardiac diseases, active or uncontrolled infections, HIV-positive patients on antiretroviral therapy, uncontrolled diabetes, cirrhosis, chronic active or persistent hepatitis, impaired respiratory function requiring oxygen-dependence, serious psychiatric disorders).
5. Pregnant or breastfeeding women.

Ages: 18 Years to 99 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 211 (Actual)
Dates: Start 2018-10-19 (Actual); Primary Completion 2025-10-17 (Actual); Study Completion 2025-10-17 (Actual)

PRIMARY OUTCOMES:
Disease Free Survival | From date of randomisation until the date of second cancer or death, which ever occurs earlier, assessed up to 5 years
  Disease free survival (DFS) defined as the time interval between randomization and physical or radiographic evidence of recurrence (local/distant) or second cancer or death (all causes) whichever occur first

SECONDARY OUTCOMES:
EORTC QLQ-C30 | through study completion, up to 2 years
  Health related quality of life of the patient
Pathological complete response (PCR) | through study completion, up to 2 years
  Pathological response will be established using the grading system called chemotherapy response score (CRS). The response will be assessed based on the omentum microscopic review.
Overall survival (OS) | from date of randomisation to death, assessed up to 5 years
  Overall survival (OS) defined as time interval between randomization and death (all causes); alive patients will be censored at the last date of news
Time for first subsequent treatment (TFST) | up to 5 years
Post-operative mortality | up to 5 months
  Post operative mortality defined as the interval between the date of debulking surgery and the date of death due to any cause occurring within the 30 day post-surgery
Post-operative morbidity | up to 5 months
  Surgical morbidity defined as the interval between the date of debulking surgery and any events occurring within the 30 day post-surgery (All grades ≥ 3 according to the CTCAE v4.03 & All grades ≥ 3 according to Clavien Dindo classification)
Fagotti laparoscopic score | diagnosis
  Disease extension assessed by Fagotti score at the time of diagnosis https://www.ncbi.nlm.nih.gov/pubmed/16791447
CTC-AE version 4.03 adverse events | 30 days after last treatment intake, up to 1 year
  safety assessment
questionnaire OV28 | through study completion, up to 2 years
  Physical, abdominal/gastrointestinal (GI), fatigue

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Marc Classe, MD, PhD, Principal Investigator — Institut de Cancérologie de l'Ouest
Locations (28):
- France (28):
  - ICA - Polyclinique Urbain V, Avignon
  - Institut Bergonié, Bordeau
  - CHU de BREST - Hôpital Cavale Blanche, Brest
  - Centre François Baclesse, Caen
  - Centre Hospitalier Universitaire Caen, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - Hôpital Simone Veil, Eaubonne
  - CHU Grenoble-Alpes - Site Nord (La Tronche), Grenoble
  - Centre Jean Bernard - Clinique Victor Hugo, Le Mans
  - CHU de Limoges - Hôpital de la Mère et de l'Enfant, Limoges
  - Hôpital du Scorff, Lorient
  - Centre Léon Bérard, Lyon
  - Hôpital Saint-Joseph, Marseille
  - ICM Val d'Aurelle, Montpellier
  - Hôpital Privé du Confluent, Nantes
  - Centre Antoine Lacassagne, Nice
  - Hôpital Cochin, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Groupe Hospitalier Pitié Salpétrière, Paris
  - Hôpital de la Milétrie - Centre Hospitalier Universitaire de Poitiers, Poitiers
  - Institut Jean Godinot, Reims
  - Hôpital René Huguenin, Institut Curie, Saint-Cloud
  - ICO Centre René Gauducheau, Saint-Herblain
  - Clinique Médico-chirurgicale CHARCOT, Sainte-Foy-lès-Lyon
  - Institut Claudius Regaud, Toulouse
  - Centre Hospitalier Universitaire Bretonneau, Tours
  - Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Classe JM, Ferron G, Ouldamer L, Gauthier T, Emambux S, Gladieff L, Dupre PF, Anota A. CHRONO: randomized trial of the CHROnology of surgery after Neoadjuvant chemotherapy for Ovarian cancer. Int J Gynecol Cancer. 2022 Aug 1;32(8):1071-1075. doi: 10.1136/ijgc-2021-003320. PMID 35321888